CLINICAL TRIAL: NCT03684928
Title: A Bilateral Dispensing Comparison of Biofinity Toric and Acuvue Vita for Astigmatism
Brief Title: A Bilateral Dispensing Comparison of Comfilcon A Over Senofilcon C Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-94
Record Dates: First submitted 2018-09-19; First posted 2018-09-26 (Actual); Results first posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2019-04

CONDITIONS: Astigmatism Bilateral

STUDY DESIGN:
Intervention Model Description: Prospective, double-masked, bilateral, randomized, one month cross-over dispensing study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Comfilcon A (test) (Active Comparator): Participants were randomized to wear either test or control contact lenses bilaterally for one month during the cross-over study.
  Interventions: Device: Comfilcon A (test); Device: Senofilcon C (control)
- Senofilcon C (control) (Active Comparator): Participants were randomized to wear either test or control contact lenses bilaterally for one month during the cross-over study.
  Interventions: Device: Comfilcon A (test); Device: Senofilcon C (control)

INTERVENTIONS:
Device: Comfilcon A (test) — Daily wear contact lenses
Device: Senofilcon C (control) — Daily wear contact lenses

SUMMARY:
The aim of this study is to evaluate the subjective acceptance of Comfilcon A contact lenses when worn on a daily wear modality over one month.

DETAILED DESCRIPTION:
This study is a 30-subjects prospective, double-masked (investigator and participant), bilateral, randomized, one month cross-over dispensing study comparing subject acceptance of Comfilcon A against Senofilcon A contact lenses.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion in the study if he/she:

1. Is at least 17 years of age and has full legal capacity to volunteer;
2. Has had a self-reported oculo-visual examination in the last two years.
3. Has read and signed an information consent letter;
4. Is willing and able to follow instructions and maintain the appointment schedule;
5. Is an adapted soft contact lens wearer, who currently wears contact lenses for a minimum 3 days/week and 8 hours/day AND who anticipates no difficulty wearing CLs for 6 days/week, 10 hours /day.
6. Is willing to wear contact lens in both eyes for the duration of the study;
7. Has a minimum astigmatism of - 0.75, determined by refraction;
8. Can be fit with the two study contact lens types in the powers available;
9. Has a distance visual acuity of 0.20 logMAR (approx 20/30) or better, determined by refraction;
10. Can achieve a distance visual acuity of 0.20 logMAR (approx 20/30) or better in each eye with the study contact lenses.
11. Has clear corneas and no active* ocular disease;

Exclusion Criteria:

A person will be excluded from the study if he/she:

1. Is participating in any concurrent clinical trial;
2. Has any known active* ocular disease and/or infection;
3. Has a systemic condition that in the opinion of the investigator may affect a study measure;
4. Is using any systemic or topical medications that in the opinion of the investigator may affect a study measure;
5. Has known sensitivity to fluorescein dye or products to be used in the study;
6. Appears to have any active* ocular pathology, ocular anomaly or severe insufficiency of lacrimal secretion (severe dry eye) that would affect the wearing of contact lenses;
7. Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit);
8. Is aphakic;
9. Has undergone refractive error surgery;
10. Has participated in the previous QUENA study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2019-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCOptom, Principal Investigator — Director, Centre for Ocular Research and Education
Locations (1):
- University Of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Comfilcon A (Test) Then Senofilcon A (Control): Participants were randomized to wear comfilcon A contact lenses first then or senofilcon C contact lenses bilaterally for one month during the cross-over study.
  Comfilcon A (test): Daily wear contact lenses
  Senofilcon C: Daily wear contact lenses
- Senofilcon C (Control) Then Comfilcon A (Test): Participants were randomized to wear Senofilcon C control contact lenses first then Comfilcon A contact lenses bilaterally for one month during the cross-over study.
  Comfilcon A (test): Daily wear contact lenses
  Senofilcon C: Daily wear contact lenses
Period: First Intervention
Arm/Group | Comfilcon A (Test) Then Senofilcon A (Control) | Senofilcon C (Control) Then Comfilcon A (Test)
Started | 23 | 22
Completed | 23 | 19
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2
Period: Second Intervention
Arm/Group | Comfilcon A (Test) Then Senofilcon A (Control) | Senofilcon C (Control) Then Comfilcon A (Test)
Started | 21 (Two participants discontinued between the first intervention and second intervention.) | 19
Completed | 20 | 19
Not Completed | 1 | 0
Not completed — Soft Tissue Injury | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Total Participants
Arm/Group | Overall Study
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.4 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 45

OUTCOME MEASURES:

1. Primary Outcome: Ease of Insertion(Handling)
Description: Subjective ratings of ease of insertion for each pair of lenses (scale: 0-10; 0= Very difficult,10 = Very easy)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Comfilcon A (Test): Participants were randomized to wear comfilcon A contact lenses bilaterally for one month during the cross-over study.
  Comfilcon A (test): Daily wear contact lenses
- Senofilcon C (Control): Participants were randomized to wear Senofilcon C control contact lenses bilaterally for one month during the cross-over study.
  Senofilcon C: Daily wear contact lenses
Arm/Group | Comfilcon A (Test) | Senofilcon C (Control)
Number analyzed (Participants) | 39 | 39
units on a scale | 9.1 (1.2) | 9.2 (1.1)

2. Primary Outcome: Ease of Insertion (Handling)
Description: Subjective ratings of ease of insertion for each pair of lenses (scale: 0-10; 0= Very difficult,10 = Very easy)
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A (Test) | Senofilcon C (Control)
Number analyzed (Participants) | 39 | 39
units on a scale | 8.9 (1.1) | 8.5 (1.9)

3. Primary Outcome: Ease of Insertion(Handling)
Description: Subjective ratings of ease of insertion for each pair of lenses (scale: 0-10; 0= Very difficult,10 = Very easy)
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Comfilcon A (Test) | Senofilcon C (Control)
Number analyzed (Participants) | 39 | 39
units on a scale | 8.8 (1.3) | 8.5 (1.7)

4. Secondary Outcome: Rotational Recovery After Lens Mislocation
Description: Lens relocation after 10 blinks, after 30º rotation mislocation
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Comfilcon A (Test) | Senofilcon C (Control)
Number analyzed (Participants) | 39 | 39
Degrees
  Nasal | 27 (4) | 23 (6)
  Temporal | 23 (8) | 19 (5)

5. Secondary Outcome: Rotational Recovery After Lens Mislocation
Description: Lens relocation after 10 blinks, after 30º rotation mislocation.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Comfilcon A (Test) | Senofilcon C (Control)
Number analyzed (Participants) | 39 | 39
Degrees
  Nasal | 26 (6) | 23 (6)
  Temporal | 23 (7) | 18 (5)

ADVERSE EVENTS:
Time Frame: From baseline up to one month for each intervention.
Arm/Group | Comfilcon A (Test) | Senofilcon C (Control)
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/28/NCT03684928/Prot_SAP_000.pdf